CLINICAL TRIAL: NCT00579696
Title: The Queens Library HealthLink Project
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other); QUEENS BOROUGH PUBLIC LIBRARY (QBPL) (Unknown); Queens Health Network (Other); Caritas Health Care, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-027
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Diseases
Keywords: Multiple Diseases; Queens

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

SUMMARY:
To determine whether community based participatory action research leads to more effective cancer prevention and control in underserved communities compared to traditional, "topdown" programs.

DETAILED DESCRIPTION:
To examine how communities engage in the participatory research process, in order to develop locally tailored initiatives for cancer education, prevention and control.

To examine whether and how long program effects are sustained after completion of the intensive collaborative program planning intervention.

ELIGIBILITY:
Inclusion Criteria:

* This project is intended to reach participants over the age of 18 within each sampled neighborhood, inclusive of both women and men of all ethnic and language groups. As such, our outcomes assessment strategy is similarly inclusive. Specific sources of data and sampling strategies for different measures are detailed in Section 7, as part of our assessment plan.

Exclusion Criteria:

* Individuals younger than 18 years of age will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Low-Income areas in the borough of Queens
Sampling Method: Non-Probability Sample
Enrollment: 2789 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To determine whether community-based participatory action research leads to more effective cancer prevention and control in underserved communities compared to traditional, "topdown" programs. | 5 years

SECONDARY OUTCOMES:
To examine how communities engage in the participatory research process, in order to develop locally tailored initiatives for cancer education, prevention and control. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Rapkin, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Web Site — http://www.mskcc.org